CLINICAL TRIAL: NCT03913026
Title: A Phase II Open-label Study of ECT-001-expanded Cord Blood Transplantation in Patients With High-risk Acute Leukemia/Myelodysplasia
Brief Title: UM171 Expanded Cord Blood In Patients With High-Risk Acute Leukemia/Myelodysplasia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Stem Cell Network (Other); ExCellThera inc. (Industry)
Responsible Party: Principal Investigator, Sandra Cohen, Associate Professor University of Montreal, Ciusss de L'Est de l'Île de Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECT-001-CB.002
Record Dates: First submitted 2019-04-09; First posted 2019-04-12 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: High Risk Hematologic Malignancy; Cord Blood Transplant
Keywords: UM171; Stem Cell Expansion
MeSH Terms: interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Main intervention (Experimental): Eligible patients will receive an ablative conditioning regimen and be infused with an ECT-001 expanded cord-blood. The ECT-001 expanded CB could be infused fresh, or cryopreserved.
  Interventions: Biological: Transplant with an expanded ECT-001 cord blood

INTERVENTIONS:
Biological: Transplant with an expanded ECT-001 cord blood — 1. Patients will receive a conditioning regimen (such as: cyclophosphamide 120 mg/kg, fludarabine 75mg/m2 and TBI 12 Gy or cyclophosphamide 50 mg/kg, fludarabine 150 mg/m2, thiotepa 10 mg/kg and TBI 4 Gy).
  2. The cord to be expanded will undergo CD34+ selection. The CD34- product is cryopreserved and will be thawed and infused on Day +1 post-transplant. The CD34+ product will be placed in a closed culture with UM171 for a 7-day expansion and is infused on Day 0.
  3. Patients will receive standard supportive care and GVHD prophylaxis (such as MMF and tacrolimus). Tacrolimus will be discontinued on Day 100 post-transplant unless GVHD arises.

SUMMARY:
Allogeneic hematopoietic stem cell transplantation is a life-saving procedure in patients with blood cancers. Cord blood (CB) represents an alternative source of stem cells, which is associated with a lower risk of relapse, especially in the presence of minimal residual disease in the setting of acute leukemia and myelodysplasia. Furthermore, CB has the added advantage of being associated with a low risk of chronic graft versus host disease (GVHD). Unfortunately, CB transplants are hampered by a higher risk of transplant related mortality (TRM) when compared to bone marrow/peripheral blood transplants because of the limited cell dose of CB.

In the previous UM171 trial (NCT02668315), the CB expansion protocol using the ECT-001-CB technology (UM171 molecule) has proven to be technically feasible and safe. UM171 expanded CB was associated with a median neutrophil recovery at day (D)+18 post transplant. Amongst 22 patients who received a single UM171 CB transplant with a median follow-up of 18 months, risk of TRM (5%) and grade 3-4 acute GVHD (10%) were low. There was no moderate-severe chronic GVHD. Thus, overall and progression free survival at 12 months were impressive at 90% and 74%, respectively. The UM171 expansion protocol allowed access to smaller, better HLA matched CBs as >80% of patients received a 6-7/8 HLA matched CB. Interestingly there were 5 patients who had already failed an allogeneic transplant and 5 patients with refractory/relapsed acute leukemia/aggressive lymphoma. Despite this high risk population, progression was 20% at 12 months. Hence, in this new trial, investigators are targeting patients with high and very high-risk acute leukemia/myelodysplasia to test the antileukemia effect of this new graft, a UM171 expanded CB.

DETAILED DESCRIPTION:
Methodology:

This is a multi-center open label phase II clinical trial. Patients with high and very high-risk acute leukemia/myelodysplasia will receive a single 5-7/8 HLA matched ECT-001 (UM171) expanded cord blood after an ablative conditioning regimen. This group of patients would be expected to have poor progression free survival (PFS) after a conventional allogeneic transplant (bone marrow-peripheral blood).

Investigators key primary and secondary objectives include:

1. To confirm low Transplant Related Mortality (TRM)
2. To evaluate relapse free survival (RFS)
3. To analyze kinetics of hematologic engraftment;
4. To evaluate the incidence of acute and chronic GVHD
5. To evaluate the safety of the procedure
6. To evaluate incidence of infectious complications
7. To analyze duration of hospitalization
8. To evaluate the incidence of pre-engraftment/engraftment syndrome (PES/ES)
9. To analyze the effect of cryopreservation of the expanded CD34+ fraction on safety and efficacy endpoints

ELIGIBILITY:
Inclusion Criteria:

1. Presence of high-risk acute leukemia/myelodysplasia defined as one of the following:

   I. Acute Myeloid Leukemia:
   1. Primary induction failure (no CR or CRi after ≥ 2 courses of induction therapy or after ≥ 1 induction containing high dose Ara-C)
   2. Chemorefractory relapse (no CR or CRi after 1 chemointensive treatment)
   3. Relapse after allogeneic or autologous transplant
   4. High risk AML in CR1: i) any adverse genetic abnormality as defined by European Leukemia Net excluding FLT3 mutation; ii) secondary or therapy related AML excluding good risk genetic abnormalities (as defined by ELN); or iii) any other poor risk feature known to be associated with a PFS or DFS ≤40% at 2 years after conventional transplantation.
   5. CR2 excluding good risk genetic abnormalities defined by ELN
   6. ≥CR3

   II. Acute Lymphoid Leukemia
   1. Primary induction failure (≥ 2 inductions)
   2. Chemorefractory relapse (at least 1 intensive induction chemotherapy; blinatumomab, inotuzumab or CAR-T cells may be considered as an equivalent)
   3. Relapse after allogeneic or autologous transplant
   4. High risk ALL in CR1: Ph like ALL or any other poor risk feature known to be associated with an PFS or DFS ≤40% at 2 years after conventional transplantation.
   5. ≥CR2
   6. MRD+ within 1 month of start of conditioning regimen.

   III. Myelodysplastic syndrome
   1. Relapse after allogeneic or autologous transplant
   2. ≥10 % blasts within 1 month of start of conditioning regimen
   3. Very poor cytogenetics (>3 abnormalities)
   4. Any poor risk feature known to be associated with a PFS or DFS ≤40% at 2 years after conventional transplantation
   5. TP53 mutation
   6. ≥40 years old and RAS or JAK2 mutation
   7. CMML with HCT-specific CPSS score high or intermediate-2
   8. Stable disease (absence of CR/PR/HI) after 6 cycles of azacitidine (or another demethylating agent)
   9. Progressive disease while on azacitidine (or another demethylating agent)
2. 18-70 years old
3. Availability of 2 CBs ≥ 4/8 HLA match when A, B, C and DRB1 are performed at the allele level.

   I. Cord to be expanded:
   1. CD34+ cell count >0.5 x 105/kg and TNC>1.5 x 107/kg (these numbers are all pre-freeze)
   2. Needs to be erythrodepleted by bank prior to cryopreservation
   3. Must come from a cord bank that is FACT (Foundation for the Accreditation of Cellular Therapy) accredited, FDA approved or eligible for NMDP IND.

   II. Non-expanded CB/back-up cord:
   1. Pre-freeze TNC count ≥ 2.0 x 107/kg with CD34+ cells ≥1.5 x 105/kg or TNC count ≥ 1.5 x 107 TNC/kg with CD34+ cells ≥1.7 x 105/kg. If a single cord does not meet these criteria, 2 back up cords will be an acceptable alternative with a minimum for each of 1.5 x 107/kg TNC and 1 x 105/kg CD34+ cells; another acceptable HSC back up source could be a haploidentical donor with medical clearance prior to starting conditioning regimen.
   2. Must come from a cord bank that is FACT accredited, FDA approved or eligible for NMDP IND
4. Karnofsky score ≥ 70%
5. Bilirubin < 2 x upper limit of normal (ULN) unless felt to be related to Gilbert's disease or hemolysis; AST and ALT ≤ 2.5 x ULN; alkaline phosphatase ≤ 5 x ULN.
6. Estimated or measured creatinine clearance ≥ 60 ml/min/1.73m2.
7. Hematopoietic cell transplantation specific comorbidity index (HCT-CI) ≤5 for patients < 60 years old; HCT-CI ≤3 for patients < 60 years old and acute leukemia not in CR/CRi; HCT-CI ≤3 for patients 60-65 years old; HCT-CI ≤1 if 66-70 years old.
8. Left ventricular ejection fraction ≥ 40%
9. Forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1) and diffusing capacity corrected for hemoglobin (DLCOc) ≥ 50% of predicted
10. Signed written informed consent
11. Female patients of childbearing potential must have a negative serum pregnancy test within 7 days of enrolment and must be willing to use an effective contraceptive method while enrolled in the study.

Exclusion Criteria:

1. Patient never treated with cytotoxic chemotherapy and planned conditioning regimen does not include 12 Gy TBI (exceptions allowed if approved by PI).
2. Allogeneic myeloablative transplant within 6 months.
3. Autologous hematopoietic stem cell transplant within 6 months.
4. Planned use of ATG in conditioning regimen (exceptions allowed if approved by PI in which case ATG must be adjusted for weight/lymphocyte count and given more than 1 week prior to transplant; any patient who receives ATG will have immune recovery studies but will not be counted with rest of patients and will be analyzed separately).
5. Planned use of an HLA matched CB (8/8 allele matched)
6. Uncontrolled infection.
7. Presence of a malignancy other than the one for which the CB transplant is being performed, with an expected survival estimated to be less than 75% at 5 years.
8. Seropositivity for HIV.
9. Hepatitis B or C infection with measurable viral load. Patients with chronic hepatitis B or C infection regardless of viral load require clear documentation of absence of cirrhosis by either fibroscan or biopsy. If fibroscan is the method used, the test must be unequivocally negative.
10. Liver cirrhosis.
11. Active central nervous system involvement
12. Chloroma > 2 cm
13. ≥50% blasts in marrow in an evaluable marrow sample (>25% of normal cellularity for age) collected less than one month prior to start of conditioning regimen.
14. Peripheral blasts >1000/mm3
15. Pregnancy, breastfeeding or unwillingness to use appropriate contraception.
16. Participation in a trial with an investigational agent within 30 days prior to entry in the study.
17. Patient unable to give informed consent or unable to comply with the treatment protocol including appropriate supportive care, follow-up, and tests.
18. Any abnormal condition or laboratory result that is considered by the PI capable of altering patient's condition or study outcome.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Transplant Related Mortality (TRM) | 1 year
  TRM is defined as any death of any cause other than malignant relapse, occurring after the commencement of conditioning regimen that could be related to the transplantation procedure.
Relapse Free survival (RFS) | 2 years
  RFS will be measured from time of transplant until disease relapse, death or last follow-up.
Overall survival (OS) | 2 years
  OS will be measured from time of transplant until disease relapse, death or last follow-up.

SECONDARY OUTCOMES:
Neutrophil Engraftment | 42 days
  Time to neutrophil engraftment is defined as the first day of attainment of an absolute neutrophil count (ANC) ≥0.5 x 109/L for 3 consecutive days. Time to ANC ≥ 0.1 x 109/L will also be documented as it seems to predict TRM.
Graft failure | 42 days
  Absence of neutrophil engraftment by day 42 or secondary graft failure without any obvious cause.
Platelet Engraftment | 60 days
  Platelet engraftment is defined as the first day of a sustained platelet count ≥ 20 x 109/L with no platelet transfusion in the preceding 7 days as per CIBMTR standards (www.cibmtr.org).
Incidence of Acute Graft Versus Host Disease (aGVHD) | 1 year
  The time to onset and maximal grade will be recorded. Acute GVHD will be defined as classic acute (time of onset of symptoms ≤ 100 days) or persistent, recurrent, or late onset acute GVHD (time of onset of symptoms > 100 days) as defined by the NIH. Results will be compared to patients at the same institution transplanted with different stem cell sources.
Incidence of Chronic Graft Versus Host Disease (cGVHD) | 2 years
  Defined as per NIH global severity scores for mild, moderate, and severe chronic GVHD.
Adverse events grade 3 or higher | 3 years
  All adverse events occurring during the clinical trial, including the protocol-defined post-treatment follow-up period, qualifying as a grade ≥ 3 toxicity per the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Incidence of severe infectious complications. | 3 years
  Any of the following infections requiring systemic therapy will be captured: invasive candidiasis, aspergillus, other invasive fungi, CMV, adenovirus, EBV, HHV-6, HSV, VZV, PCP, toxoplasmosis and mycobacterium.
Hospitalization events | 1 year
  Total number of days admitted to the hospital in the first 100 days following transplant. Last day of fever (≥38.0°C) prior to engraftment, and number of days of parenteral feeding during transplant admission.
Incidence of preengraftment/engraftment syndrome (ES) requiring therapy. | 30 days

OTHER OUTCOMES:
Immune reconstitution | 1 year
  T, B, NK cell evaluation
Identify markers suggesting escape from the immune system | 3 years
  If the underlying disease recurs, sequencing will be performed of the leukemias/MDS to identify markers suggesting escape from the immune system: for example down regulation of HLA on cancer cells.
Graft composition and evaluation | 7 days
  To better understand the effect of ECT-001 expansion a sample of the graft will be transplanted into mice before and after expansion. In addition, the different cell populations of the graft will be analyzed by flow cytometry before and after expansion. UM171 appears to increase significantly the proportion of dendritic cell precursors and mast cell precursors. Confirmation of this observation from the 1st trial will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Cohen, MD, Principal Investigator — Ciusss de L'Est de l'Île de Montréal
Locations (1):
- CIUSSS de l'Est-de-l'île-de Montreal, Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada